CLINICAL TRIAL: NCT04827615
Title: Evaluation of the Ambuja Cement Foundation Noncommunicable Disease Program in Bathinda District of Punjab, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Ambuja Cement Foundation (Unknown)
Responsible Party: Principal Investigator, Shilpa N Bhupathiraju, Assistant Professor, Department of Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB19-1217
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-05

CONDITIONS: Non Communicable Diseases; Blood Pressure; Behavior, Health; Blood Glucose, High; Blood Glucose, Low; Diabetes Type 2; Lifestyle-related Condition; Body Weight
Keywords: Evaluation; Non Communicable Disease; Body weight; Diet
MeSH Terms: conditions — Noncommunicable Diseases; Health Behavior; Diabetes Mellitus, Type 2; Mental Disorders; Body Weight

STUDY DESIGN:
Intervention Model Description: The study design is stepped wedge randomized cluster trial (4 villages in the first 6 months; additional 4 villages added every 6 months over the next 12 months) - randomized implementation.
  Staff will visit 10 target villages to screen participants for high NCD risk using Community Based Assessment Checklist scoring. For adults meeting eligibility criteria, trained enumerators will (1) complete 2 brief surveys (2) measure waist circumference (3) measure blood pressure. Follow-up visits will be scheduled to measure fasting blood glucose. For adults who meet high-risk criteria for diabetes & hypertension, an additional survey will be conducted on the 2nd day covering dietary intake & clinical history. 3 additional follow-up visits will be completed every 6 months for 18 months. Each visit will include: 2 surveys like baseline, measurements of waist circumference, blood pressure, & fasting blood glucose.
  All participants identified as high risk will be referred to a public hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Risk (Other): Group 2: Of all adults in (1), those at high risk of diabetes and hypertension, defined as having a score >4 based on the following criteria:
  * Age 40-49 years (+1), age ≥50 years (+2)
  * Used to smoke or use smokeless tobacco products or sometimes currently use (+1), currently use daily (+2)
  * Currently consume alcohol daily (+1)
  * Waist circumference 81-90 cm (women)/91-100 cm (men) (+1), >90 cm (women)/>100cm (men) (+2)
  * Physical activity <150 minutes per week (+1)
  * Parent and/or sibling with high blood pressure, diabetes, or heart disease (+2)
  Interventions: Behavioral: Ambuja Cement Foundation's Non Communicable Disease Program
- Eligible adults (Other): Group 1: All adults ≥30 years old living in the 12 target villages who meet eligibility criteria and provide informed consent
  Interventions: Behavioral: Ambuja Cement Foundation's Non Communicable Disease Program

INTERVENTIONS:
Behavioral: Ambuja Cement Foundation's Non Communicable Disease Program — Government level: Strengthening linkages with Govt; Ensuring availability & affordability of NCD diagnostics and treatment; Establishing a follow-up mechanism with patients to ensure continuity of care & medication compliance
  Provider level: Capacity building of frontline workers; Promotion of interface between community & service provider
  Community level: Screening of hypertension & diabetes for all adults ≥30 years in the village in coordination with Govt under 'population based screening'; Create awareness of modifiable risk factors and lifestyle change among high-risk population; Community mobilization & active participation in various health marker days; Formation of support groups, women's groups, self help groups, with involvement of people living with NCDs
  Individual level: Behavior change communication with messages on NCD risk factors; Nutrition awareness on healthy and unhealthy food practices

SUMMARY:
This is an academic evaluation of a program being implemented by the Ambuja Cement Foundation (ACF). The aim of the evaluation is to determine the effect of the ACF noncommunicable disease (NCD) program on (1) fasting blood glucose (a biomarker of diabetes), (2) systolic blood pressure, (3) diastolic blood pressure, and (4) body weight.

ACF will be implementing a program on NCD management. Due to resource constraints, the program will be implemented stepwise (e.g. four villages in the first 6 months then an additional four villages added every 6 months over the next 12 months). In order to improve the interpretation of the evaluation data, the team will randomize the order in which the program is implemented in the 12 villages. The design is therefore a stepped wedge randomized cluster trial. This design is ideal for (1) minimizing the practical, logistical, and financial constraints associated with large-scale project implementation, (2) control for the effect of time, and (3) ensure that all villages in the project are eventually offered the intervention.

DETAILED DESCRIPTION:
Evaluation visits will be conducted at the participant's home. At baseline, the ACF field team will first administer a screening questionnaire to all adults in the household to confirm eligibility. For those adults who meet all eligibility criteria, trained enumerators will (1) complete two brief surveys, (2) measure their waist circumference and body weight, and (3) measure their blood pressure using an automatic digital blood pressure machine. The surveys will cover demographics, family history of disease, tobacco and alcohol use, physical activity, and standard clinical symptoms. The field team will then schedule a follow-up visit within the next week to measure fasting blood glucose using a point-of-care device. For those adults who meet criteria for being high-risk for diabetes and hypertension (criteria defined further in the next section), trained enumerators will also administer an additional survey on this second day that covers dietary intake and clinical history including medication use.

For high-risk adults, after the baseline visit, three additional follow-up visits will be completed every 6 months for a total duration of 18 months. Each follow-up visit will include: two brief surveys covering the same content summarized above for baseline, as well as measurements of waist circumference, body weight, blood pressure, and fasting blood glucose. The visits will be scheduled such that participants are fasting on the day of the visit, thus allowing all visit activities to be completed in 1 day.

All surveys will be completed via interviews by trained field enumerators who will enter participant responses into password-protected tablets (Qualtrics offline mobile app).

The total population of these 12 villages is 60,701 according to the 2011 Census. All adults ≥30 years old meeting eligibility criteria will be enrolled, which is estimated to be ~40% of the total population or ~24,280 people. Based on ACF's current programming in 2 other villages in this district, it is expected that 40% of those screened (Group 1 participants) will be high-risk (Group 2 participants) or ~9,720 people (~810 per village).

For fasting blood glucose, a sample of 12 clusters in a complete stepped-wedge cluster-randomized design with 4 time periods (including the baseline), 3 steps, 4 clusters switching from control to treatment at each step, and an average of 500 participants per cluster with an average of 125 participants per cluster per time period (for a total sample size of 6000 subjects) achieves 90% power to detect a difference between means of 0.32 mmol/L (4% of anticipated mean baseline level). The test statistic used is the two-sided Wald Z-Test. The intra-class correlation coefficient (ICC) is 0.010, and the significance level of the test is 0.050. Given that near to 9000 participants are expected to be enrolled, the team is exceptionally well powered to detect significant effects in this evaluation even if there is loss to follow up.

ELIGIBILITY:
Inclusion Criteria:

* • Reside in the study area (12 villages in Bathinda District of Punjab, India). "Residence" will be defined as sleeping in a house in that village on a typical weeknight.

  * ≥30 years old. Age will be confirmed by directly viewing a government-issued document with the individual's date of birth.
  * Willing to provide informed consent.

Exclusion Criteria:

* • Plan to move permanently out of the study area in the next 12 months.

  * Pregnant (women via self-report).
  * Persons who are bedridden or mentally challenged.
  * Persons who speak a language other than Punjabi, Hindi, or English

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11322 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Glucose | Four measures over 12 months
  Fasting blood glucose will be measured using a point-of-care device
Systolic and Diastolic blood pressure | Four measures over 12 months
  Blood pressure will be measured using an automatic digital blood pressure machine
Body weight | Four measures over 12 months
  Body weight will be measured using a weighing scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ambuja Cement Foundation, Bathinda, Punjab, India